CLINICAL TRIAL: NCT06552884
Title: The Effect of Maternal Role Training Program Based on Theory on Maternal Role Attainment Mother Infant and Father Infant Attachment
Brief Title: The Effect of Maternal Role Training Program on Maternal Role Attainment Mother Infant and Father Infant Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Zeliha Karapelit, Lecturer, Amasya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 147258As.
Record Dates: First submitted 2023-09-05; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Care Pattern, Maternal
Keywords: Attachment; Maternal Role; Nursing Approach; Mercer Maternal Role Attainment Theory

STUDY DESIGN:
Intervention Model Description: After the pre-test was applied to the mother and father candidates included in the experimental group, "Maternity Identity Development Training" was given in the prenatal and postnatal period. This training program, based on Ramona T. Mercer's model of mothering role ability and covering four stages, was given to parents in their own homes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): As a nursing approach, a 4-session motherhood identity development training was given to the experimental group based on the Maternal Role Attainment Theory
  Interventions: Behavioral: (Maternity Identity Development Training)
- control group (No Intervention): Not intervention

INTERVENTIONS:
Behavioral: (Maternity Identity Development Training) — Monitoring the Effect of the Education Given to Parents According to Maternal Role Ability Theory on Maternal Role Mother-Baby and Father-Infant Attachment
  Arms: experimental group

SUMMARY:
Aim: This study was conducted to determine the effect of education prepared according to the Mother Role Attainment Theory on mothering role, mother-infant attachment,father-infant attachment Material and Method: The study was conducted with primiparous pregnant women and their spouses who applied to Amasya University Sabuncuoğlu Serefeddin Training and Research Hospital between June 2021 and May 2022 as a pretest-posttest quasi-trial model with a control group. The study was completed with 109 parents (54 experimental group, 55 control group). Introductory Information Form, Prenatal Attachment Scale, Semantic Difference Scale (Me as Mother - My Baby), Maternal Attachment Scale, Pharis Self-Confidence Scale, Prenatal Father Attachment Scale and Father-Baby Attachment Scale were used to collect data. Institutional and ethical permissions were obtained to start the research. As a nursing approach, a 4-session motherhood identity development training was given to the experimental group based on the Maternal Role Attainment Theory.Number, percentage, mean, standard deviation, chi-square dependent and independent groups t test, Mann Whitney U test and Wilcoxon sign test were used in the analysis of the data.

DETAILED DESCRIPTION:
After the pre-test was applied to the mother and father candidates included in the experimental group, "Maternity Identity Development Training" was given in the prenatal and postnatal period. This training program, based on Ramona T. Mercer's model of mothering role ability and covering four stages, was given to parents in their own homes by taking the necessary precautions, since it would be risky for the participants to be given in groups due to the COVID-19 Pandemic process. The training, which consisted of 2 sessions in the last trimester of pregnancy, 2 sessions at the end of the delivery before discharge and within the first week, and 4 sessions in total, lasted approximately 40 minutes. In addition, the parents in the training group were given a training booklet and the researcher's phone number for counseling and follow-up if needed.The training booklet, which contains the same information as the training content, was given to the parents in the experimental group at the end of the first training, and to the parents in the control group after the post-tests were administered.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate
* Being at 28-32 weeks of gestation
* Age range of 18-45
* Married and living with her spouse
* Living in the center of Amasya
* Willingness to communication and cooperation
* There is no risk in terms of maternal and fetal health.
* Not having a psychiatric health problem

Exclusion Criteria:

* Those outside the determined gestational week
* Those who are closed to communication and cooperation
* People living outside the city center of Amasya
* Those with health problems or risky pregnancies were not included in the study. Exclusion Criteria
* Loss of fetus
* Not participating/completing the trainings for any reason
* Change of residence outside the province
* Giving birth in another hospital
* Having maternal and/or newborn health problems
* To fill in the assessment tests incompletely/not at all

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — between the ages of 18-45 and 28-32 coming for antenatal follow-ups. The study consisted of primiparous pregnant women and their spouses. Although the mother and father candidates are included in the study, since the age and gestational weeks of the mother candidates have an important place in the inclusion criteria, the suitability for gender outweighs the woman.
Enrollment: 109 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Prenatal Father Attachment Scale | third trimester of pregnancy, before training
  The minimum score that can be obtained from the scale is 16, while the maximum score is 80.
  As the score obtained from the scale increases, the level of attachment also increases.
Prenatal Attachment Inventory | third trimester of pregnancy, before training
  From the scale, where the level of attachment increases as the score increases, the lowest score can be 21 and the highest score can be 84.
  As the score obtained from the scale increases, the level of attachment also increases.
Father-Baby Attachment Scale | 42nd day postpartum
  High scores indicate high levels of attachment.A high mean score is evaluated positively.Each item of the scale is scored from 1 to 5 and The lowest score that can be obtained from the scale is 19 and the highest score is 95.
  is changing
Maternal Attachment Scale | 42nd day postpartum
  It is stated that as the score obtained from the scale increases, the level of attachment also increases.A high score indicates high maternal attachment. The lowest score obtained from the scale varies between 26 and the highest score 104.
Semantic Differential Scale-Me as a Mother | third trimester of pregnancy, before training and 42nd day postpartum
  The lowest score from the scale is 11, the highest score is 77, and high scores indicate positive motherhood self-evaluation.
Semantic Differential Scale-My Baby: | third trimester of pregnancy, before training and 42nd day postpartum
  The lowest score from the "My Baby" scale is 6, the highest score is 42, and high total scores indicate the evaluation of positive baby perception.
Pharis Self-Confidence Scale | third trimester of pregnancy, before training and 42nd day postpartum
  The lowest score from the "Pharis Self-Confidence" scale is 1 and the highest score is 65, and high total score results indicate high self-confidence in baby care.

CONTACTS AND LOCATIONS:
Overall Officials: Behice Erci, professor, Study Director — Inönü University
Locations (1):
- Amasya Universty, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No